CLINICAL TRIAL: NCT05920837
Title: The Relationship Between Upper Extremity Viscoelastic Properties and Functionality in Sub-acute Stroke Patients
Brief Title: Relationship Between Upper Extremity' Viscoelastic Properties and Functionality in Subacute Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Gaziantep (Other)
Collaborators: Sanko University (Other)
Responsible Party: Principal Investigator, Ogr Uyesi Tuba MADEN, Assisstanf Profesor, University of Gaziantep
Other Study IDs: 2023/04
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Stroke; Stiffness of Right Hand, Not Elsewhere Classified; Muscle Tone Abnormalities; Functional; Bleeding
MeSH Terms: conditions — Stroke; Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke: Sample of stroke patients
  Interventions: Device: MyotonPRO; Other: Box and Block Test

INTERVENTIONS:
Device: MyotonPRO — Muscles' viscoelastic properties assess with myotonPRO.
  Other Names: Viscoelastic properties
Other: Box and Block Test — Upper extremity's functionality assess with Box and Block Test.
  Other Names: Functionality Test

SUMMARY:
In stroke patients, the shoulder-upper extremity complex is affected and reduces independence and quality in activities of daily living. Investigating the relationship between the functions of the upper extremity muscles and viscoelastic properties is important in understanding the rehabilitation of individuals with stroke.

DETAILED DESCRIPTION:
Upper extremity functions of individuals will be measured and correlated with viscoelastic properties of upper extremity muscles. The box and block test will be used for the function test. The viscoelastic properties of the muscles will be measured with the myotonPRO device. Deltoideus, Triceps, Biceps, Brachioradialis and Extansor digitorum longus were evaluated with myotonPRO. The tonus, stiffness and elasticity of muscles were recorded. Assessments will applied bilaterally and average recorded.

ELIGIBILITY:
Inclusion Criteria:

Patients who had ischemic SVO 3-9 months ago Individuals who have had a stroke for the first time MAS ≤ 2 of spasticity in paretic upper extremity

Exclusion Criteria:

TIA survivors Presence of cognitive deficits ( Mini-Mental State Examination score ≥ 24) Presence of another neurological, neuromuscular or orthopedic disease Presence of diseases that cause pain, such as fibromyalgia or arthritis Comorbidity with depression or psychiatric illness

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Individuals between the ages of 18 and 50 who had an ischemic stroke for the first time will be included in the study. Individuals with impairments that may affect upper extremity performance will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-26 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-07 (Estimated)

PRIMARY OUTCOMES:
Stiffness | through study completion, an average of one month
  stiffness (N/m) is a biomechanical feature of the muscle that characterizes its resistance to a contraction or an external force.
Elasticity | through study completion, an average of one month
  The elasticity is measured as a logarithmic decrement (log) of the natural oscillations in the tissue. Logarithmic decrement describes the tissue's ability to restore its shape after being deformed
Tone | through study completion, an average of one month
  Oscillation frequency (Hz) refers to the tone of a muscle while resting,
Functionality- Box and Block Test | through study completion, an average of one month
  Te Box and Block Test (BBT) is one of the most used and recommended tools to evaluate unilateral manual dexterity. The BBT comprises a box divided into two compartments by a wooden separation and 150 small wood cubic blocks (1-inch). The BBT consists of displacing a maximum number of small blocks, one-by-one, from the compartment located on the tested side to the other using the same hand (taking care to pass over the separation). Te score is obtained by counting the number of blocks correctly displaced within 60 s.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuba Maden, Gaziantep, Sahinbey, Turkey (Türkiye)

REFERENCES:
- [Derived] Maden T, Polat H, Guner MA, Turhan B. Alterations in proximal shoulder muscles in stroke-related pain: a myotonometric study. Ir J Med Sci. 2025 Dec;194(6):2401-2407. doi: 10.1007/s11845-025-04098-w. Epub 2025 Sep 30. PMID 41026398